CLINICAL TRIAL: NCT03059693
Title: Efficacy and Safety of HAT1, a Novel Topical Therapeutic: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Tolerability of HAT1 in Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haus Bioceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCTP16MD01
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Dermatitis, Atopic
Keywords: Eczema; Topical
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sponsor will send all washout and test products in compliance with current Good Manufacturing Practices directly to the clinical facility prior to the start of the study. Study procedures will be in place to ensure double-blind administration of study treatments. Access to the randomization code will be strictly controlled. The quantity of all study material shipped to the clinical facility will be documented on the shipping and receiving form included within the shipment. Due to the objectives of the study, the identity of test and control treatments will not be known to investigators, care provider, outcomes assessor, research staff, or patients. Packaging and labeling of test and control treatments will be identical to maintain the blind. Products will be identified with the codes generated by the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAT1 topical cream (Experimental): HAT1 medicated cream will come in a blinded tube. The research team will provide instructions for the correct application of the treatment. The medicated cream will be applied twice daily (morning and evening) at least 4 hours apart to all lesions. Treatment will continue daily until next visit. If a lesion disappears, patients will continue applying the cream twice daily to the area.
  Interventions: Drug: HAT1 topical cream
- Vehicle cream (Placebo Comparator): Vehicle cream will come in a blinded tube. The research team will provide instructions for the correct application of the treatment. The vehicle cream will be applied twice daily (morning and evening) at least 4 hours apart to all lesions. This will be continued daily until next visit.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: HAT1 topical cream
  Other Names: HAT1
  Arms: HAT1 topical cream
Drug: Vehicle cream
  Other Names: Placebo
  Arms: Vehicle cream

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory skin disease characterized by a disturbance of epidermal-barrier function that results in intensely pruritic subacute and chronic eczematous plaques. As the most common cause of chronic inflammatory skin diseases, AD is a major cause of morbidity and suffering, affecting upto 30% of children, and increasing in prevalence throughout the world. It is estimated that the direct cost of AD in the US alone ranged from $0.9 billion to $3.8 billion every year. The current therapy of AD is reactive, where the flares are treated through symptomatic management with topical corticosteroids and calcineurin inhibitors. Given that these medications have long-term side-effects, and given the chronically relapsing immunopathogenic nature of AD, there is an imperative need for safer anti-inflammatory medications. Haus Bioceuticals (Haus) has developed a topical treatment for eczema/atopic dermatitis (AD) denoted HAT1, and have demonstrated that HAT1 is safe and profoundly effective in the treatment of AD, controlling signs and symptoms in 85% of patients with AD. This study is aimed to further evaluate the potential of developing HAT1 as an integral part of AD therapy.

DETAILED DESCRIPTION:
This study is a 17 week (119 days) randomized, double-blind, in home use study among 48 male and female subjects with moderate to severe active atopic dermatitis (AD). The study will include subjects with ages 12 - 65 years old inclusive. Group assignments will be balanced by disease severity, age, and body location of AD lesions (listed in order of importance). The study will consist of a 1 week washout period, 12 week treatment phase and a 4 week regression phase. During the treatment phase, subject will be provided one of the two test products to use twice daily on all lesions and non-lesional areas as instructed. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study. Measurements, expert visual assessments and self-assessments will be taken as described below. Safety and tolerability will be evaluated by incidence of AE's (defined per CTCAE), exacerbations, application site reactions/infections, and lab evals. There will also be consumption/compliance checks and dermatological evaluations at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe atopic dermatitis as determined by Physician's Global Assessment (PGA > 3)
* Males and females, age 12 - 65 years old inclusive

Exclusion Criteria:

* Is currently participating or has participated in another interventional clinical study at this or any other facility in the past 2 weeks.
* Currently or has been diagnosed or treated for cancer in the past 5 years.
* Requires any topical or systemic medications that could affect the course of their atopic dermatitis during the study period (except inhaled steroids and/or stable antihistamines for asthma or allergies).
* Has a known hypersensitivity to any corticosteroid creams.
* Has any active infections or has used antibiotics in the past 7 days.
* Has any physical attributes or skin conditions that might interfere with the clear visual or instrumental assessments.(i.e. cuts, sunburn, birth marks, tattoos, extensive scarring, excessive hair growth or acne)
* Has an immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus rheumatoid arthritis) which could place the subject at risk or interfere with the accuracy of the study results.
* Has used any immunosuppressant drugs or immunotherapy within the past 30 days or 5 half-lives.
* Is an employee of the sponsor company or clinical testing site.
* Is dependent on oral medication for any skin disease/condition or could not, in the opinion of the Investigator tolerate the restriction of discontinuing the medicine as required in this study.
* Is currently pregnant or lactating or planning to become pregnant in the next 6 months (using double contraception for prevention).
* Has a history of keloid formation following skin injury.
* Is routinely taking anti-coagulant medications (i.e. Plavix, Coumadin, warfarin, heparin, etc.)
* Any other condition or factor the Investigator or their duly assigned representative believes may affect the ability of the subject to complete the study or the interpretation of the results.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2016-07-24 (Actual)

PRIMARY OUTCOMES:
Change in Scoring of Atopic Dermatitis (SCORAD) score | Baseline to week 12

SECONDARY OUTCOMES:
Absolute change in Eczema Area and Severity Index (EASI) score | Baseline to week 12
Proportion of patients achieving a Physician's Global Assessment (PGA) score of 0 or 1 | Baseline to week 12
Incidence of treatment emergent AE's | Baseline to week 12

IPD SHARING:
Plan to Share IPD: Yes